CLINICAL TRIAL: NCT00195559
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of a Combination of Levonorgestrel and Ethinyl Estradiol in a Continuous Daily Regimen in Subjects With Premenstrual Dysphoric Disorder
Brief Title: Study Evaluating Combination of Levonorgestrel and Ethinyl Estradiol in Pre-Menstrual Dysphoric Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0858A4-318
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Premenstrual Syndrome; Menstruation Disturbances
Keywords: Premenstrual Syndrome (PMS); Hormone Therapy
MeSH Terms: conditions — Premenstrual Syndrome; Menstruation Disturbances | interventions — Ethinyl Estradiol-Norgestrel Combination

INTERVENTIONS:
Drug: Levonorgestrel/Ethinyl Estradiol

SUMMARY:
The purpose of this study is to determine whether Levonorgestrel/Ethinyl Estradiol (LNG/EE) is effective in treating the symptoms of severe Premenstrual Dysphoric Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, women aged 18 to 49 years.
* History of severe PMS symptoms over the last year, as determined by the investigator.
* Regular 21 to 35 day menstrual cycle for 2 months prior to first study visit.

Exclusion Criteria:

* Major depressive disorder requiring antidepressant treatment or hospitalization within the last 3 years.
* Contraindication to combination oral contraceptives.
* Use of antidepressants/anxiolytics within 10 days of screening and for the duration of the study.

Other exclusion applies.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 526 (Estimated)
Dates: Start 2005-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Mean change in average Daily Record of Severity of Problems (DRSP) 21-item total daily score

SECONDARY OUTCOMES:
Change from baseline in DRSP 21-item daily score based on the 5 days with the highest DRSP scores in each "estimated" treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Trial Manager, Principal Investigator — For Argentina, Chile, scheima@wyeth.com; Trial Manager, Principal Investigator — For Brazil, xavierl@wyeth.com; Trial Manager, Principal Investigator — For Denmark, Finland, Sweden, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Germany, MedinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Mexico, gomezlj@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Managersp, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Romania, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For UK, ukmedinfo@wyeth.com
Locations (51):
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Rosario-Santa Fe
- Brazil (6):
  - Curitiba
  - Goiânia
  - Porto Alegre
  - Salvador
  - São Paulo
  - Sorocaba
- Chile (2):
  - Santiago
  - Temuco
- Denmark (4):
  - Aarhus
  - Frederiksberg
  - København NV
  - Rungsted Kyst
- Finland (4):
  - Helsinki
  - Kuopio
  - Oulu
  - Turku
- Germany (4):
  - Berlin
  - Bonn
  - Hamburg
  - Hanover
- Mexico (6):
  - Lomas de Virreyes, D.F.
  - Guadalajara, Jalisco
  - Zapopan, Jalisco
  - Monterrey, N.L.
  - San Luis Potosí City, San Luis Potosí
  - Mexico City
- Netherlands (5):
  - Amsterdam
  - Apeldoorn
  - Den Helder
  - Enschede
  - Nieuwegein
- Poland (5):
  - Bialystok
  - Gdansk
  - Mysłowice
  - Poznan
  - Warsaw
- Romania (3):
  - S, Bucharest
  - Cluj-Napoca
  - Iași
- Sweden (4):
  - Gothenburg
  - Stockholm
  - Umeå
  - Uppsala
- United Kingdom (5):
  - Conwell
  - Fowey
  - London
  - Plymouth
  - St Austell